CLINICAL TRIAL: NCT05369611
Title: COVID-19 Experiences in the SELF Cohort: A Cross-Sectional Study
Brief Title: COVID-19 Experiences in the SELF Cohort
Status: Enrolling by invitation | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000811; 000811-E
Record Dates: First submitted 2022-05-07; First posted 2022-05-11 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-03-21

CONDITIONS: COVID-19
Keywords: Fibroid; Natural History
MeSH Terms: conditions — COVID-19; Leiomyoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SELF: 1,668 current members of the SELF cohort: African American women between the ages of 23-35 at enrollment in SELF who have not previously withdrawn from SELF and are not known to have died.

SUMMARY:
Background:

COVID-19 affected African Americans more than Whites. African Americans, especially women, have had higher rates of COVID-19 infections compared to Whites. They are also more likely to go to the hospital or die of this disease. Many researchers who looked into these issues lacked background data on the people they studied. SELF is a 10-year study of fibroids in African American women aged 23-35. Researchers already have a lot of data on these women. Asking how COVID-19 affected them can add context other studies lack.

Objective:

To describe the impact of the COVID-19 pandemic on young African American women and their families.

Eligibility:

Participants must be enrolled in SELF (Study of Environment, Lifestyle, and Fibroids).

Design:

Researchers will invite all women enrolled in SELF to participate in this natural history study.

Participants will complete one questionnaire. They will answer the questions online. They may also choose to get a paper copy sent by mail. The survey will take no more than 15-20 minutes.

All questions will relate to COVID-19. Participants will be asked if they had COVID-19. They will be asked if family, friends, or members of their community did. They will answer questions about their vaccine status and access to health care services.

Participants will also answer questions about how the pandemic affected their lives. They will be asked about their job and if finding childcare was a challenge. They will be asked about money problems and how they coped. They will be asked about sleep problems and emotional distress.

Participants will get a $30 gift card after they finish the survey.

DETAILED DESCRIPTION:
Study Description:

This cross-sectional study will be an add-on to the Study of Environment, Lifestyle and Fibroids (SELF) (Protocol Number: 10-E-N044). SELF is a prospective cohort study of fibroid development. From November 2010 to December 2012, the study enrolled a volunteer sample recruited from Detroit, MI and surrounding areas of approximately 1,700 African-American women ages 23-35 without a diagnosis of fibroids. SELF has been a rich information source regarding the health of young African-American women.

This current COVID-19 study will focus on collecting information regarding SELF participant s experiences throughout the COVID-19 pandemic through a short, one-time online questionnaire. The questionnaire will contain questions on a range of topics related to the COVID-19 pandemic to include 1) pandemic experiences in the following domains: COVID-19 illness of participant (including LONG-COVID), participant s family and friends, participants social community 2) vaccination status, 3) access to health care, 4) employment vulnerabilities and employment loss, 5) challenges with caring for children, 6) financial hardship, coping strategies, 7) sleep problems, and 8) psychosocial stressors. The questionnaire will also ask questions about COVID-19-related symptoms, vaccination, and hospitalizations experienced by the participants and/or members of her household and community.

Objectives:

Primary Objective:

To describe the impact of the COVID-19 pandemic on reproductive-aged African American women and their families. We have three goals:

First, these basic data will be summarized in a report that will be sent back to the participants. Like our newsletters, this will serve as a cohort maintenance activity, keeping our participants interested and engaged in the study.

Secondly, SELF collaborators are continuing to follow the participants (the 4th follow-up is in progress, and a 5th follow-up is being planned), so these data will allow us to consider the impact of COVID-19 in future analyses. Additional studies with this cohort could also be undertaken in the future. Depending upon the exposure outcome being investigated in the data from those additional follow ups, an overall measure of impact may be important, or the impact on specific domains may be of most interest.

Thirdly, we also view this study as an opportunity to document the impact of the COVID-19 pandemic, a once in a century event, in a well characterized group of reproductive-aged African-American women whose health and well-being have been followed for nearly a decade now. This is an understudied group and documenting their response to COVID will serve as one of several case-studies of specific subpopulations that are likely to emerge after the pandemic. The goal is to document the range of adverse impacts experienced and the factors (e.g., low income, limited educational attainment, pre-pandemic health conditions, neighborhood factors) that might mitigate or exacerbate those adverse impacts for this understudied demographic group.

Endpoints:

Primary Endpoint: Descriptive data on impact of the COVID-19 pandemic on reproductive-aged African American women and their families

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Ongoing enrollment in the NIEHS s Study of Environment, Lifestyle & Fibroids (SELF) cohort (i.e. not deceased or previously withdrawn from SELF)
* Ability to complete the questionnaire (indicating informed consent)

EXCLUSION CRITERIA:

-Not enrolled in the NIEHS the NIEHS s Study of Environment, Lifestyle & Fibroids (SELF) cohort (i.e. not deceased or previously withdrawn from SELF)

Ages: 23 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will be the 1,668 current members of the SELF (10E0044) cohort. These are African American women who were between the ages of 23-35 at enrollment in SELF who, to date, have not previously withdrawn from SELF and are not known to have died
Sampling Method: Non-Probability Sample
Enrollment: 1668 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
COVID-19 | 24 months
  Primary Endpoint: Descriptive data on impact of the COVID-19 pandemic on reproductive-aged African American women and their families

CONTACTS AND LOCATIONS:
Overall Officials: Chandra L Jackson, Ph.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- National Institute of Environmental Health Sciences (NIEHS), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided